CLINICAL TRIAL: NCT00001265
Title: Studies on the Natural History and Pathogenesis of Polymyositis, Dermatomyositis, and Related Diseases
Brief Title: Study and Treatment of Inflammatory Muscle Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910196; 91-AR-0196
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: Autoimmune Diseases; Idiopathic Inflammatory Myopathies; Dermatomyositis; Inclusion Body Myositis; Pathogenesis; Natural History; Connective Tissue Diseases
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Autoimmune Diseases; Myositis; Myositis, Inclusion Body; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Patients with no disease
- Patients with muscle disease: Patients with known or suspected Idiopathic Inflammatory myopathies (IIM)

SUMMARY:
This study of inflammatory muscle diseases-polymyositis and dermatomyositis and related disorders-will examine what causes these diseases and describe the clinical features (signs and symptoms) associated with them. Inflammation and degeneration of skeletal muscles in these disorders leads to weakness and muscle wasting. The skin, lungs and other organs may also be involved.

Patients 16 years of age and older with polymyositis, dermatomyositis, or a related disorder may be eligible for this study. Participants will undergo a complete history and physical examination, including routine blood and urine tests. Additional procedures for diagnosis, treatment or research may include:

1. Blood sample for genetic studies.
2. Muscle biopsy-removal of a tissue sample for microscopic examination. Under local anesthetic, a 1/2- to 1-inch long incision is made in the thigh or upper arm, and a small piece of muscle is removed.
3. Electromyography-measurement of the electrical activity of a muscle. A needle is inserted through the skin into a muscle to record its electrical activity.
4. Magnetic resonance imaging-visualization of organs or tissues, using a magnetic field and radio waves. The patient lies on a table inside a narrow cylinder (the MRI scanner) with a strong magnetic field for the scanning.
5. Manual muscle strength testing by a physiotherapist.
6. Swallowing studies using ultrasound (imaging using sound waves) and X-rays (barium swallow) to evaluate swallowing and speaking abilities.
7. Questionnaires on swallowing ability and ability to perform daily living activities
8. Pulmonary function tests-measurement of movement of air in and out of the lungs. The patient breathes into a machine to evaluate lung function.
9. Chest X-rays to evaluate lung function.
10. Electrocardiogram and, if necessary, Holter monitoring (measurement of the electrical activity of the heart) and echocardiogram (ultrasound imaging of the heart) to evaluate heart function.
11. Apheresis-collection of white blood cells for research. Whole blood is collected through a needle placed in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are removed and the rest of the blood is returned to the body through the same needle or through a second one placed in the other arm.
12. MR guided muscle biopsy-measurement of glycogen in muscle tissue using magnetic resonance imaging. Certain patients may undergo this experimental procedure to compare MRI findings with those of muscle biopsy. The affected muscles are identified using MRI and the biopsy incision is made. MRI is then used to guide the biopsy needle to the muscle and a small piece is removed.

Patients who are eligible for experimental treatment studies will be offered the opportunity to join them. Others will be advised of treatment recommendations.

DETAILED DESCRIPTION:
Polymyositis, dermatomyositis and related disorders, also known as the idiopathic inflammatory myopathies (IIM), are an uncommon, heterogeneous group of diseases. This is an omnibus protocol designed to continue our description of this rare group of diseases, further delineate important groups of patients, and obtain useful material for further study of immunological abnormalities, pathogenesis and etiology of IIM. Often the diagnosis of an IIM can be confused with other illness (such as adult-onset dystrophies), and therefore, we will be evaluating patients with other illnesses (who are referred with a preliminary diagnosis of an IIM) (1). Patients evaluated with IIM will receive (with informed consent) the best standard therapies available and consideration for entry into any therapeutic protocols. MRI will be performed on healthy volunteers to help develop a mathematical method for quantitating edema of muscle MRI in patients (2). MRI/PET will be performed on some patients and on healthy volunteers to evaluate its role in understanding muscle disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

All eligible patients are invited to participate in this protocol. Patients are adults and minors, aged 16 or higher, with possible idiopathic muscle disease (suspected or confirmed). Since both men and women are affected with the disease, both sexes will be studied. All ethnic and racial groups are at risk and will be included. Pregnant women and women who intend to become pregnant during the study will be eligible since this disease affects both segments of the population. This protocol proposes responsible inclusion of pregnant women and the justification for this derives in part from the fact that women (who are suffering from autoimmune and rheumatic diseases) lack data from which to make informed decisions about health care during pregnancy.

INCLUSION OF PREGNANT WOMEN:

The majority of patients with autoimmune disease are women and of these individuals, the majority are of childbearing age. Furthermore, pregnancy is a risk factor for fluctuations in autoimmune disease activity, including organ- and life- threatening flares. The majority of our study population is comprised of women. The exclusion of women who become pregnant from systemic study by way of our natural history protocol, threatens both the well-being of the individual women (owing to the standard of care provision of the protocol) and the systematic discovery of pregnancy-specific data concerning the immunopathological basis of autoimmune disease. Skewed understanding from a restricted natural history study may leave vulnerable groups open to disproportionate harm owing to inequities in research. In other words, automatic disqualification due to pregnancy denies women agency in the issue of gender equity for access to research and in addition the systematic exclusion of pregnant women prevents generalizability of information to help under-resourced and marginalized populations, nationwide.

In summary,

* The cost of exclusion of pregnant women with myositis 1) insufficient evidence concerning how to manage such disease for the population, and 2) lack of access to the best myositis specific advice for individuals enrolled in the protocol who are unlikely to have access to specialty care outside of the NIH
* The cost of exclusion in research with regard to fetal safety derives from the fact that preeclampsia, eclampsia, preterm birth and miscarriage are higher in women who do not have access to subspecialty care. In this situation, reticence on the part of nonspecialists to treat active autoimmune disease during pregnancy or lack of access to appropriate treatment may lead to harm to women and their fetuses.
* The pregnant body possesses a unique hormonal and immunological environment. Similarly, it metabolizes medications in a manner different from non-pregnant women, let alone men. Hence, there is no reasonable path towards generating important biomedical knowledge other than to include pregnant women in this protocol.

The tension between protection by exclusion and the presumption of inclusion in research protocols has been specifically addressed by the US Institute of Medicine (now National Academy of Medicine) and the Task Force on Research Specific to Pregnant Women and Lactating Women to advise the Secretary of Health and Human Services regarding gaps in knowledge and research on safe and effective therapies for pregnant and lactating women, and both have both weighed in as favoring the presumption of inclusion (https://www.nichd.nih.gov/about/advisory/PRGLAC). Our study falls in line with these position papers since it is responsible (it benefits, patients and their fetuses and provides relevant data to the population at large) and because it is low risk (it is standard of care, only, and does not invoke experimental interventions).

Healthy volunteers will be eligible only if they are adults aged 18 or older and only if they are willing to provide informed consent. There is no benefit to the healthy volunteers; however their inclusion will provide invaluable information in comparison to the patients for the purpose of research. Recruitment of healthy volunteers has been completed.

Participation of NIH Staff or family members of study team members

NIH staff and family members of study team members may be enrolled in this study as this population meets the study entry criteria. Neither participation nor refusal to participate as a subject in the research will have an effect, either beneficial or adverse, on the participant s employment or position at NIH.

Every effort will be made to protect participant information, but such information may be available in medical records and may be available to authorized users outside of the study team in both an identifiable an unidentifiable manner.

The NIH Information Sheet on NIH Staff Research Participation will be made available. Please see section for consent of NIH Staff.

EXCLUSION CRITERIA:

* Children (age less than 16 years) are excluded
* Subjects with severe active infection (such as requiring intravenous antibiotics) or other co-morbidities that in the opinion of the investigator would warrant exclusion.
* Subjects or their legal guardians who are unable or unwilling to give informed consent/assent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Volunteers and patients with known or suspected Idiopathic Inflammatory myopathies (IIM)
Sampling Method: Non-Probability Sample
Enrollment: 1325 (Actual)
Dates: Start 1992-01-10 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Muscle strength | End of Study
  To determine its utility in differentiating different muscle diseases, in identifying early extra muscular involvement of muscle diseases, in characterizing the pattern of muscle involvement for the diseases studied, and whether it can serve as a diagnostic tool to better identify muscle inflammation and atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Mammen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.At this time, It is not yet known if there will be a plan to make IPD available . The protocol is silent about IPD sharing.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1991-AR-0196.html